CLINICAL TRIAL: NCT04795973
Title: Effects of Intermittent Fasting on Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Guang Wang, Head of the Endocrinology Department, Beijing Chao Yang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2021-IF-11
Record Dates: First submitted 2021-03-10; First posted 2021-03-12 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Sensitivity to Thyroid Hormones; Metabolic Parameters; in Patients With FLD
Keywords: fatty liver disease; 5:2 intermittent fasting; thyroid hormone sensitivity; insulin sensitivity; weight loss
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Insulin Resistance; Weight Loss

STUDY DESIGN:
Intervention Model Description: Inclusion criteria were hepatic fat content (HFC) > 5.0% evaluated by upper abdominal MRI proton density fat fraction (MRI-PDFF) examinations, age ≥ 18 years, body mass index (BMI) ≥ 18.5 kg/m2, and stable body weight (change < ± 10% of body weight) during the last 3 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 5:2 intermittent fasting (Experimental): All subjects received 5:2 IF. They followed a normal diet for 5 days each week and practiced IF for 2 days discontinuously. On normal eating days, women consumed 1200 to 1500 kcal/day and men consumed 1500 to 1800 kcal/day, with macro-nutrient distribution of 45% to 50% carbohydrate, 20% protein, and 30% to 35% fat. They consumed 500 kcal and at least 50 g of protein on a light fasting day. Noncaloric beverages like water and unsweetened tea were allowed without restriction. A nutritionist provided diet guidance and documented any discomfort symptoms throughout the study.
  Interventions: Behavioral: 5:2 intermittent fasting

INTERVENTIONS:
Behavioral: 5:2 intermittent fasting — All subjects received 5:2 IF. They followed a normal diet for 5 days each week and practiced IF for 2 days discontinuously. On normal eating days, women consumed 1200 to 1500 kcal/day and men consumed 1500 to 1800 kcal/day, with macro-nutrient distribution of 45% to 50% carbohydrate, 20% protein, and 30% to 35% fat. They consumed 500 kcal and at least 50 g of protein on a light fasting day. Noncaloric beverages like water and unsweetened tea were allowed without restriction. A nutritionist provided diet guidance and documented any discomfort symptoms throughout the study.

SUMMARY:
Eighty subjects with FLD were recruited from the endocrinology clinic at Beijing Chao-yang Hospital. All of the following inclusion criteria needed to be met: hepatic fat content (HFC) were upper 5.0% evaluated by upper abdominal MRI proton density fat fraction (MRI-PDFF) examinations, age ≥ 18 years, body mass index (BMI) ≥ 18.5 kg/m2, and stable body weight (change < ± 10% of body weight) during the last 3 months. Participants underwent an 8-week 5:2 IF intervention. Metabolic parameters and thyroid hormone sensitivity indices were assessed at baseline and after intervention.

DETAILED DESCRIPTION:
Eighty subjects with FLD were recruited from the endocrinology clinic at Beijing Chao-yang Hospital, Capital Medical University, China, between September 22, 2020 and April 30, 2021. Inclusion criteria were hepatic fat content (HFC) > 5.0% evaluated by upper abdominal MRI proton density fat fraction (MRI-PDFF) examinations, age ≥ 18 years, body mass index (BMI) ≥ 18.5 kg/m2, and stable body weight (change < ± 10% of body weight) during the last 3 months. Participants underwent an 8-week 5:2 IF intervention. Metabolic parameters and thyroid hormone sensitivity indices were assessed at baseline and after intervention.

ELIGIBILITY:
Inclusion Criteria:

* hepatic fat content (HFC) > 5.0% evaluated by upper abdominal MRI proton density fat fraction (MRI-PDFF) examinations
* age ≥ 18 years
* body mass index (BMI) ≥ 18.5 kg/m2
* stable body weight (change < ± 10% of body weight) during the last 3 months

Exclusion Criteria:

* plasma aspartate aminotransferase (AST) and alanine amino-transferase (ALT) levels exceeded 2.5 times of the upper limit of normal
* fasting blood glucose (FBG) levels ≥ 7.0 mmol/L or glycated hemoglobin A1c (HbA1c) ≥ 6.5%
* with type 1 or type 2 diabetes
* with heart disease
* with other hepatic disease (excluding FLD)
* with renal disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (BMI, kg/m²) measured using digital scale and stadiometer | 8 weeks
  BMI will be calculated as weight (kg) divided by height squared (m²). Weight will be measured on a calibrated digital scale and height using a stadiometer. Measurements will be taken at baseline and after the 8-week intermittent fasting intervention.
TSH Index (TSHI) calculated from serum TSH and FT4 levels | 8 weeks
  Fasting venous blood samples will be collected at baseline and after the 8-week intermittent fasting intervention. Serum TSH and FT4 concentrations will be determined using a standardized automated immunoassay. TSH Index will be calculated according to published formulas.
Thyrotroph Thyroid Hormone Sensitivity Index (TTSI) calculated from serum TSH and FT4 levels | 8 weeks
  Fasting blood samples will be collected at baseline and after the 8-week intermittent fasting intervention. Serum TSH and FT4 concentrations will be measured using a standardized automated immunoassay. TTSI will be calculated according to published formulas.
FT3/FT4 ratio calculated from serum FT3 and FT4 levels | 8 weeks
  Fasting venous blood samples will be collected at baseline and after the 8-week intermittent fasting intervention. Serum FT3 and FT4 concentrations will be measured using a standardized automated immunoassay, and the FT3/FT4 ratio will be calculated as an index of peripheral thyroid hormone conversion efficiency.
Changes in metabolic parameters after 8-week IF intervention, measured using blood tests and biochemical assays. | 8 weeks
  Lipid profile: Total cholesterol (TC), triglycerides (TG), low-density lipoprotein cholesterol (LDL-C), and high-density lipoprotein cholesterol (HDL-C) will be measured from fasting blood samples.
  Glycated hemoglobin (HbA1c, %) will be measured using high-performance liquid chromatography (HPLC). Fasting glucose (mg/dL or mmol/L) will be measured using an enzymatic glucose oxidase method. Fasting insulin (μIU/mL) will be measured using an electrochemiluminescence immunoassay. All blood samples will be collected after an overnight fast at baseline and after the 8-week IF intervention.
Changes in abdominal MRI findings (liver fat deposition) after 8-week IF intervention, assessed using magnetic resonance imaging | 8 weeks
  Abdominal fat distribution and liver fat content will be assessed using magnetic resonance imaging (MRI). Scans will be performed at baseline and after the 8-week IF intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Guang Wang, Principal Investigator — Beijing Chao-Yang Hospital, Capital Medical University, Beijing 100020, China
Locations (1):
- Beijing Chao-yang Hospital, Capital Medical University, Beijing, Beijing Municipality, China